CLINICAL TRIAL: NCT03990727
Title: Phenotype Correlates Genotype of Inherited Retina Dystrophies
Brief Title: Phenotype Correlates Genotype of Inherited Retina Dystrophies, Retinitis Pigmentosa, Con>Rod Dystrophies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MejoraVisionMD (Network)
Collaborators: Maisonneuve-Rosemont Hospital (Other); Retina and Genomics Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: RETMxMap
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Retinitis Pigmentosa; Cone Dystrophy; Usher Syndromes; Retina; Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Cone Dystrophy; Usher Syndromes; Retinal Dystrophies | interventions — Optical Imaging; Genotype

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Retinitis pigmentosa: Any type of retina dystrophy with pigment / retinitis pigmentosa
  Interventions: Diagnostic Test: Retina Analysis-mosaic; Diagnostic Test: Autofluorescence; Diagnostic Test: OCT- 1 micra; Procedure: Genotype analysis
- Usher Syndrome: Retina dystrophy or retinitis pigmentosa associated with audition problems
  Interventions: Diagnostic Test: Retina Analysis-mosaic; Diagnostic Test: Autofluorescence; Diagnostic Test: OCT- 1 micra; Procedure: Genotype analysis
- Cone>rod syndromes: Retina dystrophy diagnosed or started in central vision.
  Interventions: Diagnostic Test: Retina Analysis-mosaic; Diagnostic Test: Autofluorescence; Diagnostic Test: OCT- 1 micra; Procedure: Genotype analysis
- Retinitis pigmentosa sx: Retinitis pigmentosa with any type of other features
  Interventions: Diagnostic Test: Retina Analysis-mosaic; Diagnostic Test: Autofluorescence; Diagnostic Test: OCT- 1 micra; Procedure: Genotype analysis

INTERVENTIONS:
Diagnostic Test: Retina Analysis-mosaic — Fundus retina pattern study
Diagnostic Test: Autofluorescence — Fundus reflectance-functionality
Diagnostic Test: OCT- 1 micra — Fine tomography fundus retina
Procedure: Genotype analysis — Molecular target retina dystrophy analysis

SUMMARY:
Patients with retina dystrophies (retinitis pigmentosa, cone>rods dystrophies, Usher and syndromic) will be correlated with genotype and validate inheritance mode by segregation analysis.

DETAILED DESCRIPTION:
Patients with retina dystrophies (retinitis pigmentosa, cone>rods dystrophies, Usher and syndromic, etc.) will be correlated with genotype and validate inheritance mode by segregation analysis. Ocular exam of proband, parents and two unaffected siblings is needed, retina analysis, autofluorescence and ocular coherence tomography (OCT) are needed as well as family map. Blood samples 10ml max blood extraction will be sent and genotype will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of inherited retina dystrophy or retinitis pigmentosa
2. Must be able to perform all study tests.
3. Must be able to visit every year.

Exclusion Criteria:

1) Not willing to visit every year.

Ages: 2 Weeks to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inherited retina dystrophies / Retinitis pigmentosa, LCA, Cone-rod dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Estimated)
Dates: Start 2009-08 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Gene-molecular variation to correlate with phenotype based on autofluorescence, retina analysis, | 8 years
  Molecular variation correlates with specific phenotype based on autofluorescence, retina analysis, macular coherence tomography.

SECONDARY OUTCOMES:
Preliminary Natural History | 5 years
  Ocular exam, retina analysis, autofluorescence and OCTs will be described in time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Retina and Genomics Institute, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
It will be share by publication papers.
Supporting Information: SAP, CSR
Time Frame: 1a
Access Criteria: To organism with known knowledge in the field. To expand analysis in same field. Via digital, by contacting administrator.
URL: http://mejoravisionmd.com

REFERENCES:
- [Result] Villanueva, Adda L., et al.
- [Result] Villanueva, A. L., Langlois, M., Mongrain, I., Provost, S., Asselin, G., Dubé, M. P., ... & Ayyagari, R. (2015). ARRP microarray and Exome analysis revealed known and novel mutations in Mexican pedigrees. Investigative Ophthalmology & Visual Science, 56(7), 2866-2866.